CLINICAL TRIAL: NCT01575236
Title: A Randomized Non Crossover Study of the GuardianTM Versus SupremeTM Laryngeal Mask Airway
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Schulthess Klinik (Other)
Collaborators: Medical University Innsbruck (Other)
Responsible Party: Principal Investigator, ChristianKeller, MD, M.Sc., Schulthess Klinik
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Schulthess_Anä_3; Schulthess_Anä_3 (Other: Schulthess Klinik)
Record Dates: First submitted 2012-03-30; First posted 2012-04-11 (Estimated); Last update posted 2012-08-08 (Estimated); Status verified 2012-08

CONDITIONS: Adverse Anesthesia Outcome

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Guardian (Experimental): Guardian Laryngeal Mask
  Interventions: Device: Guardian Laryngeal Mask
- Supreme (Experimental): Supreme Laryngeal Mask Airway
  Interventions: Device: Supreme Laryngeal Mask Airway

INTERVENTIONS:
Device: Guardian Laryngeal Mask — ease of insertion, oropharyngeal seal pressure, fiberoptic position, ease of ventilation, occult blood, gastric insertion
  Other Names: Guardian Laryngeal Mask, Umedaes
  Arms: Guardian
Device: Supreme Laryngeal Mask Airway — ease of insertion, oropharyngeal seal pressure, fiberoptic position, ease of ventilation, occult blood, gastric insertion
  Other Names: Supreme Laryngeal Mask Airway, LMA Deutschland GmbH
  Arms: Supreme

SUMMARY:
The investigators test the hypothesis that ease of insertion, oropharyngeal leak pressure, fiberoptic position and ease of gastric tube placement differ between the GuardianTM and the LMA SupremeTM in paralyzed, anesthetized patients.

DETAILED DESCRIPTION:
The GuardianTM is a new extraglottic airway device which brings together features of both the LMA ProSealTM (high seal cuff, gastric access and bite block - to facilitate ventilation, airway protection and airway obstruction, respectively) and the LMA UniqueTM (single use - prevention of disease transmission). In the following randomized, non-crossover study, the investigators test the hypothesis that ease of insertion, oropharyngeal leak pressure, fiberoptic position and ease of gastric tube placement differ between the GuardianTM and the LMA SupremeTM in paralyzed, anesthetized patients.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1 or 2
* Age 18-75 yr
* Written informed consent

Exclusion Criteria:

* Difficult airway
* Non fasted
* BMI > 35

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2012-03; Primary Completion 2012-06 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
efficacy of oropharyngeal seal pressure | 5 min
  this will be measured over the full range of cuff volumes (0-40 ml) and at an intracuff pressure of 60 cm H2O

SECONDARY OUTCOMES:
anatomic position | 5 min
  this will be determined fiberoptically via the airway tube over the full range of cuff volumes and at an intracuff pressure of 60 cm H2O

CONTACTS AND LOCATIONS:
Overall Officials: Christian Keller, MD MSc, Study Chair — Anästhesie Schulthess Klinik
Locations (1):
- Universitätsklinik für Anästhesie, Innsbruck, Tyrol, Austria